CLINICAL TRIAL: NCT07221240
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Amisodin in Healthy Adult Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Amisodin in Healthy Adult Subjects With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PRG Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PRG-A-001
Record Dates: First submitted 2025-09-30; First posted 2025-10-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: The study includes SAD, MAD and a food effect cohort. While the overall study uses a parallel design, the food effect cohort is conducted using a crossover design.
Who Masked: Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Amisodin (Experimental): Subjects who have successfully completed the screening phase will enter the treatment phase of the study and be randomized to a treatment arm. Subjects randomized to the Amisodin arm will receive orally administered Amisodin either as a single ascending dose (SAD) or multiple ascending doses (MAD) under fasting conditions, with one cohort in the SAD part crossing over to receive the same dose under fed conditions to assess the effect of food.
  Interventions: Drug: Amisodin
- Drug: Placebo (Placebo Comparator): Subjects who have successfully completed the screening phase will enter the treatment phase of the study and be randomized to a Placebo arm. Subjects randomized to the Placebo arm will receive orally administered Placebo either as a single ascending dose (SAD) or multiple ascending doses (MAD) under fasting conditions.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amisodin — Administered as specified in the treatment arm.
  Arms: Drug: Amisodin
Other: Placebo — Administered as specified in the Placebo arm.
  Arms: Drug: Placebo

SUMMARY:
Researchers will evaluate the safety, tolerability, and pharmacokinetics (PK) of orally administered Amisodin in healthy adult subjects through a randomized, double-blind, placebo-controlled Phase 1 study consisting of two parts: single ascending dose (SAD) and multiple ascending dose (MAD). The food effect will be assessed in one cohort in Part1. Approximately 32 healthy, adult subjects are planned to be enrolled in total. Subjects will participate in only one part and one cohort.

DETAILED DESCRIPTION:
During this trial, a total of 32 subjects will be randomized in a 3:1 ratio (out of 8 subjects, 6 on Amisodin, 2 on placebo in each dose group). The placebo is a capsule that looks like Amisodin but contains no study drug. The use of a placebo helps to make sure that any side effects during the study are judged fairly.

In Part 1 (SAD), subjects will receive a single oral dose of Amisodin or placebo under fasting conditions, with one cohort crossing over to receive the same treatment under fed conditions to assess the effect of food. In Part 2 (MAD), subjects will receive Amisodin or placebo once daily for 7 days under fasting conditions. Dose escalation in both parts will proceed only after safety and tolerability are confirmed by the Safety Review Committee (SRC). Safety assessments will include adverse events (AEs), ECGs, vital signs, laboratory tests, physical examinations, and C-SSRS evaluations, while plasma samples will be collected to evaluate PK.

Amisodin will be administered study drug or placebo with approximately 180mL of water under fasting conditions. The capsules will be opened and mixed with 60mL of water. The contents will be stirred well to create a uniform suspension for consumption and immediately administered orally as one dose to the subject. The cup/bottle will be rinsed with an additional 60mL of water and immediately administered to the subject. A second rinse with an additional 60mL of water will be performed and immediately administered to the subject.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

* 1. Healthy, adult, male or female (of non-childbearing potential only)*, 18 55 years of age, inclusive, at the screening visit.

  * Females of non-childbearing potential are defined as follows:

    * Females who have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

      o Hysteroscopic sterilization

      o Bilateral tubal ligation or bilateral salpingectomy

      o Hysterectomy
      * Bilateral oophorectomy or
    * Females who are postmenopausal with amenorrhea for at least 1 year prior to the first dosing and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status. 2. Male subjects must follow protocol specified contraception guidance as described in Section 7.4.5 Contraception Requirements and agree to refrain from sperm donation until 90 days after the last dosing. 3. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing based on subject self-reporting.

      4. Body mass index (BMI) ≥ 18.0 and < 32.0 kg/m2 at the screening visit. 5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, or vital signs, as deemed by the PI or designee at the screening visit, including the following:
    * Seated blood pressure is ≥ 90/50 mmHg and ≤ 140/90 mmHg
    * Liver function tests at or below limit or normal range
    * Estimated glomerular filtration rate (estimated by Modification of Diet in Renal Disease Study equation [MDRD] method) ≥ 90 mL/min/1.73 m² 6. No ECG findings of clinical significance as judged by the PI or qualified designee at the screening visit and at first check in, including each criterion as listed below:
    * Normal sinus rhythm (heart rate between 40 and 100 bpm, inclusive)
    * QTcF interval ≤ 450 msec (males) or ≤ 460 msec (females)
    * QRS interval < 110 msec; if > 110 msec, result will be confirmed by a manual over read
    * PR interval ≤ 210 msec 7. Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

* 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.

  2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee. 3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study. 4. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing. 5. History or presence of hypersensitivity or idiosyncratic reaction to compounds related to the study drug, study drug excipients, or antihistamines.

  6. Allergy to band aids, adhesive dressing, or medical tape. 7. Female subjects of childbearing potential. 8. Female subject with a positive pregnancy test at the screening visit or at first check-in or who is lactating. 9. Positive urine drug or serum alcohol results at the screening visit or first check-in. 10. Positive results at the screening visit for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV). 11. Unable to refrain from or anticipates the use of:

  • Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing.

  • Any drugs known to be significant inducers of cytochrome P450s (CYP) and/or P-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first dosing.

  • Any drugs that prolong the QT/QTc interval within 14 days (or 5 half lives, whichever is longer) prior to the first dosing.

  12. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing. 13. Donation of blood or significant blood loss within 56 days prior to the first dosing. 14. Plasma donation within 7 days prior to the first dosing 15. Participation in another clinical study within 90 days prior to the first dosing.

The 90-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.

16. Any other reason determined by the PI or designee, in their opinion, that would prevent the subject's participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Number and severity of TEAEs following a single oral dose of Amisodin and placebo. | From signing of the informed consent form until the follow-up visit (7 days [± 1 day] after dosing).
  To evaluate the safety and tolerability of a single ascending dose of Amisodin in healthy adult subjects.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4 MAD- Day 1
  AUC0-t-The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4
  AUC0-inf -The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4
  AUC%extrap -Percent of AUC0-inf extrapolated, represented as (1 - AUC-t/AUC-inf) ×100.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4
  CL/F - Apparent total plasma clearance after oral (extravascular) administration, calculated as Dose/AUC0-inf.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4 MAD- Day 1
  Cmax-Maximum observed concentration.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4 MAD- Day 1
  Tmax -Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4
  Tlag-Lag time- the delay between study drug administration and the onset of absorption (applicable to FE Cohort S2 only).
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4 MAD- Day 7
  Kel -Apparent first-order terminal elimination rate constant calculated from a semi log plot of the plasma concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero plasma concentrations).
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4 MAD- Day 7
  t1/2 -Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel.
Pharmacokinetics (PK) of Amisodin | SAD- Day 1 to Day 4
  Vz/F -Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration, calculated as Dose/(AUC0-inf × Kel).
Pharmacokinetics (PK) of Amisodin | MAD- Day 1 to Day 7
  Ctrough-Plasma trough concentration observed at the end of the dosing interval
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  AUCtau -The area under the concentration-time curve during a dosing interval (tau) at steady state.
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  Cmax,ss-Maximum observed concentration at steady state.
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  Cmin,ss-Minimum observed/measured non-zero concentration at steady state.
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  Tmax,ss-Time to reach Cmax,ss over the final dosing interval. If the maximum value occurs at more than one time point, Tmax,ss is defined as the first time point with this value.
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  CLss/F-Apparent total plasma clearance at steady state after oral (extravascular) administration, calculated as Dose/AUCtau.
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  Cavg-Average plasma concentration during the dosing interval (Ratio of AUCtau to the dosing interval, tau).
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  Vz,ss/F-Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration, calculated as Dose/(AUCtau × Kel).
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  RA_AUC Accumulation ratio calculated from AUCtau at steady-state and AUC0-t, following a single dose on Day 1. If AUC0-12 on Day 1 cannot be estimated, then corresponding AUC0-t values on Days 1 and 10 will be used instead (will be calculated where applicable).
Pharmacokinetics (PK) of Amisodin | MAD- Day 7
  RA_Cmax-Accumulation ratio calculated from Cmax,ss at steady-state and Cmax following a single dose on Day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No